CLINICAL TRIAL: NCT05928624
Title: Wireless Automated Tracking in Cirrhosis Patients at Home (WATCH) Trial: A Randomized Single Blind Trial Testing the Use of Home Monitoring Among Decompensated Cirrhosis Patients
Brief Title: A Pilot Trial to Test the Feasibility of Utilizing Home Blood Pressure Monitoring to Optimize the Administration of Midodrine Among Decompensated Cirrhosis Patients
Acronym: WATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-36046
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis, Liver; Portal Hypertension; Ascites Hepatic
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Weights and Measures; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Sham Comparator): This arm will receive a home blood pressure monitor and scale; however, these data will not be shared with their treating provider in real-time.
  Interventions: Other: Standard of Care
- Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions (Experimental): This arm will receive a home blood pressure monitor and scale. These data will be reviewed weekly and these data will be shared with the treating provider to inform clinical decisions.
  Interventions: Device: Withings Home Blood Pressure Device and Scale

INTERVENTIONS:
Device: Withings Home Blood Pressure Device and Scale — The intervention will be whether the data generated from home monitoring devices are shared with the clinical providers. The investigators are not testing the efficacy of these approved devices.
  Arms: Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions
Other: Standard of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
This is a randomized single-blind feasibility trial to test the utilization of home blood pressure devices to improve the clinical management of decompensated cirrhosis patients.

DETAILED DESCRIPTION:
This is a feasibility trial to determine the feasibility of using home monitoring devices (e.g. blood pressure cuffs) to improve outcomes for cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will need to have decompensated cirrhosis defined as a Child Pugh Score ≥ 7

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cullaro, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions
Started | 34 | 35
Completed | 34 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (2) | 61 (3) | 62 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 6 | 12
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mean Arterial Pressure (MAP) in mmHg [Mean (Standard Deviation); unit: mmHg] | 75 (5) | 77 (6) | 76 (5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Pressure
Description: The investigators will compare the change in mean arterial pressure before and after utilization of the data generated from the home monitoring.
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard of Care | Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions
Number analyzed (Participants) | 34 | 35
mmHg | 0.5 (3.2) | 1 (4.1)

2. Secondary Outcome: Change in Ascites Burden
Description: The investigators will compare the change in ascites burden, defined as the total volume of ascites removed during the study period, before and after utilization of the data generated from the home monitoring.
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Standard of Care | Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions
Number analyzed (Participants) | 34 | 35
L | 6.1 (4.2) | 4.7 (5.1)

ADVERSE EVENTS:
Time Frame: These were measured over the study period, 24 weeks.
Arm/Group | Standard of Care | Home Blood Pressure and Scale Monitoring to Inform Clinical Decisions
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT05928624/Prot_SAP_000.pdf